CLINICAL TRIAL: NCT05531656
Title: Synaptic Therapy Alzheimer's Research Trial (START): A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Trial to Evaluate the Safety and Efficacy of CT1812 in Early Alzheimer's Disease Over 18 Months.
Brief Title: A Study to Evaluate the Safety and Efficacy of CT1812 in Early Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cognition Therapeutics (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Alzheimer's Clinical Trials Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COG0203; R01AG065248 (NIH)
Record Dates: First submitted 2022-08-08; First posted 2022-09-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-07

CONDITIONS: Early Alzheimer's Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- CT1812 100 mg (Active Comparator): CT1812 at a dose of 100 n=180 group
  Interventions: Drug: CT1812
- CT1812 200 mg (Active Comparator): CT1812 at a dose of 300mg, n=180 group
  Interventions: Drug: CT1812
- Placebo (Placebo Comparator): Placebo, n=180 group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CT1812 — Study Drug
  Other Names: Study Drug Active
  Arms: CT1812 100 mg; CT1812 200 mg
Drug: Placebo — Non-active study drug
  Other Names: Matching Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter randomized, double-blind, placebo-controlled Phase 2 study designed to evaluate the efficacy, safety, and tolerability of two doses of CT1812 compared to placebo in participants diagnosed with early Alzheimer's disease.

DETAILED DESCRIPTION:
This is a multicenter randomized, double-blind, placebo-controlled Phase 2 study designed to evaluate the efficacy, safety, and tolerability of two doses of CT1812 compared to placebo for approximately 18 months (72 weeks) in approximately 540 participants diagnosed with early Alzheimer's disease

Participants will be randomized 1:1:1 to receive either 100mg or 200mg of CT1812 or placebo. CT1812 or placebo will be administered as 2 capsules to be taken orally once daily.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 50-85 years.
2. Diagnosis of either MCI due to AD or mild AD dementia.
3. MMSE 20-30 (inclusive).
4. Amyloid PET scan of the brain or CSF biomarkers consistent with AD.
5. Neuroimaging (MRI) obtained during screening consistent with the clinical diagnosis of Alzheimer's disease, as based on central read.

Exclusion Criteria:

1. Screening MRI of the brain indicative of significant abnormality.
2. Clinically significant abnormalities in screening laboratory tests.
3. Clinical or laboratory findings consistent with:

   1. Other primary degenerative dementia, (dementia with Lewy bodies, fronto-temporal dementia, Huntington's disease, Creutzfeldt-Jakob Disease, Down syndrome, etc.).
   2. Other neurodegenerative condition (Parkinson's disease, amyotrophic lateral sclerosis, etc.).
   3. Other infectious, metabolic or systemic diseases affecting the central nervous system (syphilis, present hypothyroidism, present vitamin B12, other laboratory values etc.)
4. A participant known to be actively infected with hepatitis B or hepatitis C at screening. History of acute/chronic hepatitis B or C and/or carriers of hepatitis B (seropositive for hepatitis B surface antigen [HbsAg] or anti-hepatitis C [HCV] antibody). Participants who have evidence of resolved hepatitis infection (e.g., HCV RNA negative) may be considered following discussion with the Medical Monitor.
5. A current DSM-V diagnosis of active major depression or GDS > 6, schizophrenia, or bipolar disorder.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) scale. | 18 months
  The Clinical Dementia Rating (CDR) is a clinical scale that describes 5 levels of impairment in performance on each of 6 categories of function including memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. The ratings of degree of impairment obtained on each of the 6 categories of function are synthesized into 1 global rating of dementia as absent, questionable, mild, moderate, or severe (global CDR scores of 0, 0.5, 1, 2, or 3, respectively). The score is based on interviews with the participant and study partner, using a structured interview. A sum of boxes score (CDR-SB) provides an additional measure of change where each category has a maximum possible score of 3 points and the total score is a sum of the category scores giving a total possible score of 0 to 18 with higher scores indicating more impairment.

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognition (ADAS-Cog 13) | 18 months
  Change from baseline in the Alzheimer's Disease Assessment Scale-Cognition (ADAS-Cog 13) at 18 months.
Alzheimer's Disease Cooperative Study - Activities of Daily Living Scale (ADCS - ADL) in people with Mild Cognitive Impairment (MCI) - ADCS-ADL-MCI. | 18 months
  Change from baseline in the Alzheimer's Disease Cooperative Study - Activities of Daily Living Scale (ADCS - ADL) in people with Mild Cognitive Impairment (MCI) - ADCS-ADL-MCI at 18 months.
Cerebrospinal fluid (CSF) concentrations of beta-amyloid (Aβ) 40 and 42, tau, phospho-tau (ptau), neurofilament light (NfL), neurogranin, and synaptotagmin. | 18 months
  Change from baseline at 18 months.
Plasma measures of Aβ fragments, ptau, and Neurofilament light (NfL) | 18 months
  Change from baseline at 18 months.
Volumetric Magnetic Resonance Imaging (MRI) including hippocampal and whole brain volume change | 18 months
  Change from baseline at 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Caggiano, MD, Study Director — Cognition Therapeutics
Locations (49):
- United States (49):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of California, Irvine, California
  - Stanford University, Palo Alto, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Yale University, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Mayo Clinic,Jacksonville, Jacksonville, Florida
  - JEM Research Institute, Lake Worth, Florida
  - K2 Medical Research, LLC, Maitland, Florida
  - Advanced Clinical Research Network, Corp, Miami, Florida
  - Charter Research, Orlando, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Brain Matters Research Stuart, Stuart, Florida
  - University of South Florida, Tampa, Florida
  - Conquest Research, LLC, Winter Park, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Sanders-Brown Center on Aging, Lexington, Kentucky
  - John Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Highlands Research Eastern MA, Plymouth, Massachusetts
  - University of Michigan, Ann Arbor, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University / University Hospitals, Beachwood, Ohio
  - Ohio State University, Columbus, Ohio
  - Central States Research, LLC, Tulsa, Oklahoma
  - Summit Headlands LLC, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - Ralph H. Johnson VA MC, Charleston, South Carolina
  - Vanderbilt University Medical Center Center for Cognitive Medicine, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No